CLINICAL TRIAL: NCT03787901
Title: The Ongoing Pregnancy Rate for Vitrification of Day-4 Morula and Day-5 Blastocyst
Brief Title: Comparing the Ongoing Pregnancy Rate for Vitrification of Day-4 Morula With Day-5 Blast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to achieve sample size due to COVID19 pandemic
Sponsor: Egyptian Foundation of Reproductive Endocrinology (Other)
Collaborators: Al Hayat ICSI Centre of Alexandria, Egypt (Unknown); Agial IVF/ICSI Unit of Alexandria, Egypt (Unknown); Al Madina Fertility centre of Alexandria, Egypt (Unknown); Rahem Fertility Center of Zagazig, Egypt (Unknown)
Responsible Party: Principal Investigator, Hassan Maghraby, MD, Director, Al Hayat ICSI Centre of Alexandria, Egypt, Egyptian Foundation of Reproductive Endocrinology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EFRE Vitrification Trial
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morula Vitrification Arm (Experimental)
  Interventions: Other: Morula Vitrification
- Blastocyst Vitrification Arm (Active Comparator)
  Interventions: Other: Morula Vitrification

INTERVENTIONS:
Other: Morula Vitrification — Evaluating the ongoing pregnancy rate following Morula vitrification compared with Blastocyst Vitrification.

SUMMARY:
Comparing the vitrification at Day-4 (morula stage) with the blastocyst stage vitrification outcomes with the transfer of all day 5 after warming seems need evaluation. To the best of our knowledge, there has been no random-controlled trial conducted such comparison. Altogether, this trial is to evaluate the morula stage vitrification to blastocyst vitrification on the ongoing pregnancy rate after ICSI.

DETAILED DESCRIPTION:
Vitrification of human embryos has been a paradigm-shifting procedure for higher survival rate compared with the slow freezing protocol. The evidence is scarce to support superior results for vitrifying certain stages of preimplantation embryos. Anecdotal evidence suggests that blastocyst vitrification is more forgiving than cleavage stages. However, data obtained from the procedure of assisted shrinkage of blastocysts before vitrification show a higher survival rate, suggesting that fluid accumulation insides the blastocyst can be a barrier for cryoprotectant to reach the cells. Although reassuring, whether facilitating the cryoprotectants transfer to cells by the laser-assisted shrinkage or other modalities is completely safe remains elusive. Moreover, other claims compare between day-3 embryos vitrification and blastocyst stage, suggesting no difference exists.

One of the most critical stages in embryo development is the maternal to zygotic genome activation (MZA), which occurs at the 4 to 8 cell stages. Therefore, it seems the morula stage is still cleavage but passed the MZA. Morula in the most grading system has compaction for all or the majority of cells so if vitrified, the morula stage can bypass the earlier stage of vitrification as well as the need for the artificial shrinkage for blastocyst stage. Therefore, comparing the vitrification at Day-4 (morula stage) with the blastocyst stage vitrification outcomes with the transfer of all day 5 after warming seems need evaluation. To the best of our knowledge, there has been no random-controlled trial conducted such comparison. Altogether, this trial is to evaluate the morula stage vitrification to blastocyst vitrification on the ongoing pregnancy rate after ICSI.

ELIGIBILITY:
Inclusion Criteria:

1. Women age of ≥ 18 to ≤ 40
2. BMI of ≤ 31
3. Normal responder (≥ 12 antral follicle count (AFC) during basal ultrasound examination) or hyper responder
4. The freeze-all groups including PCOS, OHSS, or high Progesterone at trigger day
5. Women who have ≥ 1 year of primary or secondary infertility
6. Tubal factor (unilateral, bilateral obstruction or salpingectomy)
7. Fresh semen ejaculates but not frozen or surgically retrieved sperm
8. Male factor: oligoasthenozoospermia but not globozoospermia or pinhead sperm
9. Women who are undergoing their first or second ICSI attempts with a previously successful attempt
10. Women who undergo only freeze-all embryo
11. Freeze-all for poor endometrium at the fresh cycle
12. Freeze-all due to abnormal endometrial findings such as polyp or myoma with a decision for freeze all for surgical correction.
13. Women who have normal endometrial thickness (≥ 8) and echo-pattern at the time of progesterone start in the proposed vitrified warmed cycle

Exclusion Criteria:

1. Women who have uncorrectable uterine pathology or abnormality including submucous myoma
2. Women or their husbands who have abnormal karyotyping
3. Women with a history of recurrent abortions or repeated implantation failures
4. Women who have uncontrolled diabetes
5. Women with diagnosed or undiagnosed liver or renal disease
6. Women who had a history of malignancy or borderline pathology
7. Women who will not meet the inclusion criteria
8. Women who will refuse to participate in the study
9. Women with endometriosis
10. Patient undergoing PGS or PGD
11. Surgically retrieved, frozen-thawed and pinpoint sperm or globozoospermia
12. Adenomyosis
13. Severe medical condition

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
The ongoing pregnancy rate | 12 weeks
  Continued pregnancy at > gestational week 12 or more per initiated cycle

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 14 days
  positive b-hCG at ≥ 14 days following embryo transfer per initiated cycle
Implantation rate | 12 weeks
  Sacs with a heartbeat on ultrasound per embryo transferred
Cumulative implantation rate | One year
  Sacs with a heartbeat on ultrasound per embryo transferred within one year from randomization
Clinical pregnancy rate | 7 weeks
  Sacs with a positive heartbeat on ultrasound at ≥ 7 weeks of gestation per initiated cycle
Cumulative clinical pregnancy rate | One year
  Sacs with a positive heartbeat on ultrasound at ≥ 7 weeks of gestation per initiated cycle within one year from randomization
Cumulative ongoing pregnancy rate | One year
  continued pregnancy after gestational week 12 per initiated cycle within one year from randomization
Twin pregnancy rate | One year
  ≥ two foetuses with a heartbeat per initiated cycle
Embryo survival rate after thawing | Five days of culture
  Blastocyst re-expansion for day 5 vitrified embryo after two hours and blastocyst formation on day 5 for embryo vitrified on day 4

CONTACTS AND LOCATIONS:
Locations (4):
- Egypt (4):
  - Agial, Alexandria
  - Al Hayat ICSI Centre of Alexandria, Alexandria
  - AlMadina IVF and ICSI Centre, Alexandria
  - Rahem Fertility Centre of Zagazig, Zagazig

IPD SHARING:
Plan to Share IPD: No